CLINICAL TRIAL: NCT04828135
Title: Characterizing the Long-Term Cardiopulmonary Effects of COVID-19 With Hyperpolarized Xenon and Cardiac MRI
Brief Title: Dual MRI for Cardiopulmonary COVID-19 Long Haulers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bastiaan Driehuys (Other)
Responsible Party: Sponsor-Investigator, Bastiaan Driehuys, Associate Professor of Radiology, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00107681
Record Dates: First submitted 2021-03-11; First posted 2021-04-01 (Actual); Results first posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Covid19
Keywords: MRI; Hyperpolarized 129Xe
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This will be a single-blinded open-label study enrolling 30 subjects (accrued 23 subjects (13 subjects who continue to have respiratory symptoms and 10 subjects within competitive sports) with a laboratory-confirmed diagnosis of COIVD-19 infection, and after 60 days or longer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- subjects with diagnosis of COVID-19 (Long-hauler) (Experimental): 23 subjects with a confirmed diagnosis of COVID-19 infection, and after 60 days or longer
  Interventions: Drug: Hyperpolarized 129Xenon gas

INTERVENTIONS:
Drug: Hyperpolarized 129Xenon gas — Each xenon dose will be limited to a volume less than 25% of subject lung capacity (TLC),
  Other Names: Xe MRI

SUMMARY:
The next phase of the COVID-19 pandemic is likely to see a surge in an associated chronic cardiopulmonary disease that will challenge health systems. Recovered patients are presenting with persistent dyspnea at the Duke Pulmonary Post-COVID clinic. Evidence is now mounting that recovered patients have significant residual pulmonary disease, while myocardial injury has also been increasingly reported. To optimally care for these patients, Duke Pulmonary study team must comprehensively assess and monitor the changes in cardiopulmonary function and relate the changes to physiologic and quality of life outcomes. The study team will deploy cutting-edge MRI to fully characterize cardiopulmonary function in enrolled 30 subjects (accrual 23 subjects) at time point 60-120 days post recovery and 6-9 months later. Cardiac MRI will assess the myocardial status and right ventricular function, while hyperpolarized 129Xe MRI will provide a 3D assessment of pulmonary ventilation, interstitial barrier integrity, and pulmonary vascular hemodynamics. The overall objective outlined in this study is to demonstrate the feasibility and value of comprehensive longitudinal imaging characterization of cardiopulmonary structure and function in patients recovered from Covid-19.

DETAILED DESCRIPTION:
The proposed research builds on the established sensitivity of Hyperpolarized 129Xe MRI to obstructive and pulmonary vascular lung disease, features expected to represented in the Covid-19 cohort. It further incorporates a new understanding of the possible role of myocardial injury in these recovered patients by combining cutting-edge pulmonary and cardiac MRI.

Although the initial presentation of patients with moderate to severe symptoms of COVID19 infections is dominated by respiratory symptoms, 10% go on to develop persistent post-infection symptoms which are thought to have an inflammatory etiology. Evidence suggests that pathologic activation of the inflammasome persists beyond the acute initial presentation that contributes to the persistent disabling symptoms characterized as "long-haul COVID". For this trial, subjects will be eligible for enrollment if subjects are outpatients with a history of a laboratory-confirmed diagnosis of COVID-19 infection, and after 60 days or longer. The study team will accrual 13 subjects who continue to have respiratory symptoms (i.e., cough, shortness of breath, dyspnea on exertion). An additional 10 subjects engaged in competitive sports and diagnosed with COVID-19 will also be enrolled. These subjects can be asymptomatic or mildly to moderately. Although rare, cardiac impairment has been documented in <2% of these individuals. The study team knowledge, XeMRI has not yet been studied in this specific patient subset.

Existing data highlight significant racial and ethnic disparities with historically underserved minority populations (i.e., Black, LatinX) suffering disproportionately higher infection rates and more severe illness compared to Whites. This is reflected by the population enrolled in the study team RedCAP database and biorepository. As such 30% of subjects enrolled will be required to be from underserved communities.

ELIGIBILITY:
Diagnosis of post Coronavirus (COVID-19)

Inclusion Criteria:

1. Age ≥ 18-year-old
2. Tested positive for SARS-CoV2
3. Willing and able to give informed consent and adhere to visit/protocol scheduled (consent must be given before any study procedures are performed)

Exclusion Criteria:

1. Prisoners
2. Pregnant, planning pregnancy, or lactating
3. Conditions that prohibit MRI scanning (metal in eye, claustrophobia, inability to lie supine).
4. Medical or psychological conditions which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Loretta Que, MD, Principal Investigator — Duke University
Locations (1):
- Duke Asthma, Allergy, and Airway Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Historical Controls were not considered enrolled.
Groups:
- Participants With Diagnosis of COVID-19 (Long-hauler): Participants with a confirmed diagnosis of COVID-19 infection, and after 60 days or longer
  Hyperpolarized 129Xenon gas: Each xenon dose will be limited to a volume less than 25% of subject lung capacity (TLC),
Period: Overall Study
Arm/Group | Participants With Diagnosis of COVID-19 (Long-hauler)
Started | 18
Completed | 13
Not Completed | 5

BASELINE CHARACTERISTICS:
Groups:
- Participants With Diagnosis of COVID-19 (Long-hauler): 23 participants with a confirmed diagnosis of COVID-19 infection, and after 60 days or longer
  Hyperpolarized 129Xenon gas: Each xenon dose will be limited to a volume less than 25% of subject lung capacity (TLC),
- Historical Controls: 10 participants with historical Hyperpolarized 129Xenon imaging
- Total: Total of all reporting groups
Arm/Group | Participants With Diagnosis of COVID-19 (Long-hauler) | Historical Controls | Total
Number analyzed (Participants) | 18 | 10 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 10 | 25
  >=65 years | 3 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 10 | 5 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 14 | 8 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 18 | 10 | 28

OUTCOME MEASURES:

1. Primary Outcome: Red Blood Cell to Membrane (RBC:M) Ratio
Description: To determine cardiopulmonary structure-function abnormalities that characterize early phase COVID-19 recovery.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: ratio (RBC:M)
Groups:
- Subjects With Diagnosis of COVID-19 (Long-hauler): Participants with a confirmed diagnosis of COVID-19 infection, and after 60 days or longer
  Hyperpolarized 129Xenon gas: Each xenon dose will be limited to a volume less than 25% of subject lung capacity (TLC),
- Historical Controls: Participants with no diagnosis of COVID-19 infection
Arm/Group | Subjects With Diagnosis of COVID-19 (Long-hauler) | Historical Controls
Number analyzed (Participants) | 13 | 10
ratio (RBC:M) | 0.39 (0.14) | 0.51 (0.13)

2. Primary Outcome: Ventilation Defect Percent
Description: To determine cardiopulmonary structure-function abnormalities that characterize early phase COVID-19 recovery.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: percentage of ventilation defect
Arm/Group | Subjects With Diagnosis of COVID-19 (Long-hauler) | Historical Controls
Number analyzed (Participants) | 13 | 10
percentage of ventilation defect | 2.4 (3.5) | 0.6 (0.7)

3. Primary Outcome: High Membrane Percent
Description: To determine cardiopulmonary structure-function abnormalities that characterize early phase COVID-19 recovery.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: percentage of high membrane
Arm/Group | Subjects With Diagnosis of COVID-19 (Long-hauler) | Historical Controls
Number analyzed (Participants) | 13 | 10
percentage of high membrane | 18.23 (29.4) | 0.5 (1.3)

4. Primary Outcome: Red Blood Cell (RBC) Defect Percent
Description: To determine cardiopulmonary structure-function abnormalities that characterize early phase COVID-19 recovery.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: percentage of RBC defect
Arm/Group | Subjects With Diagnosis of COVID-19 (Long-hauler) | Historical Controls
Number analyzed (Participants) | 13 | 10
percentage of RBC defect | 10.6 (5.6) | 4.2 (4.8)

5. Primary Outcome: Red Blood Cell to Membrane (RBC:M) Ratio at 9 Months
Description: To characterize the evolution of cardiopulmonary abnormalities over 9 months.
Time Frame: 9 Months
Measure: Mean (Standard Deviation); unit: ratio (RBC:M)
Arm/Group | Subjects With Diagnosis of COVID-19 (Long-hauler)
Number analyzed (Participants) | 13
ratio (RBC:M) | 0.44 (0.14)

6. Primary Outcome: Ventilation Defect Percent at 9 Months
Description: To characterize the evolution of cardiopulmonary abnormalities over 9 months.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: percentage of ventilation defect
Arm/Group | Subjects With Diagnosis of COVID-19 (Long-hauler)
Number analyzed (Participants) | 13
percentage of ventilation defect | 0.5 (0.5)

7. Primary Outcome: High Membrane Percent at 9 Months
Description: To characterize the evolution of cardiopulmonary abnormalities over 9 months.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: percentage of high membrane
Arm/Group | Subjects With Diagnosis of COVID-19 (Long-hauler)
Number analyzed (Participants) | 13
percentage of high membrane | 15 (30.6)

8. Primary Outcome: Red Blood Cell (RBC) Defect Percent at 9 Months
Description: To characterize the evolution of cardiopulmonary abnormalities over 9 months.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: percentage of RBC defect
Arm/Group | Subjects With Diagnosis of COVID-19 (Long-hauler)
Number analyzed (Participants) | 13
percentage of RBC defect | 6.2 (1.8)

9. Primary Outcome: Identify MRI Features That Predict Physiological Outcomes With DLCO (Diffusing Capacity of the Lungs for Carbon Monoxide)
Description: DLCO is the extent to which oxygen passes from the air sacs of the lungs into the blood.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage of predicted value
Arm/Group | Subjects With Diagnosis of COVID-19 (Long-hauler)
Number analyzed (Participants) | 13
percentage of predicted value | 20 (8)

ADVERSE EVENTS:
Time Frame: 9 Months
Description: Historical Controls were not monitored/assessed for deaths and/or adverse events.
Groups:
- Participants With Diagnosis of COVID-19 (Long-hauler): Participants with a confirmed diagnosis of COVID-19 infection, and after 60 days or longer
  Hyperpolarized 129Xenon gas: Each xenon dose will be limited to a volume less than 25% of subject lung capacity (TLC)
Arm/Group | Participants With Diagnosis of COVID-19 (Long-hauler)
All-Cause Mortality (participants affected / at risk) | 1/18
Serious Adverse Events (participants affected / at risk) | 3/18
Other Adverse Events (participants affected / at risk) | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Diagnosis of COVID-19 (Long-hauler) (N=18)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
(Respiratory, thoracic and mediastinal disorders) | 1 (1) — Adverse event is unknown; not related to the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-26): https://cdn.clinicaltrials.gov/large-docs/35/NCT04828135/Prot_SAP_000.pdf